CLINICAL TRIAL: NCT06673771
Title: Effects of Vestibular Rehabilitation on Balance and Post Stroke Fatigue: a Randomized Control Trial
Brief Title: Effects of Vestibular Rehabilitation on Balance and Post Stroke Fatigue :
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Zil-e-huma
Record Dates: First submitted 2024-11-03; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Stroke Patients
Keywords: conventional treatment; VRT Treatment; stroke population

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vestibular Rehabiliation Therapy (Experimental): VRT include head and body movemnt, eye movement, balance training
  Interventions: Other: Vestibular Rehabiliation Therapy
- Conventional Treatment (Active Comparator): conventional treatment include balance, walking, weight shifting and muscle strengthening training
  Interventions: Other: Conventional treatment

INTERVENTIONS:
Other: Vestibular Rehabiliation Therapy — Moving the eye horizontally between two stationary target while keeping the head still Moving the eye vertically between two stationary target while keeping the head still Moving the target horizontally and tracking it with the eye while keeping the head still Moving the target vertically and tracking it with the eye while keeping the head still Moving the head horizontally while a keeping a look on stationary target Moving the head vertically while a keeping a look on stationary target Moving the head and target in opposite direction horizontally while tracking the target with eyes Moving the head and target in opposite direction vertically while tracking the target with eyes.
  Sit down and stand up, sit down and stand up with eye open and eye close Stand up, but turn to the right while standing Stand up, but turn to the left while standing Place an object on the floor. Take it and bring it above your head and place it on the floor again
  Arms: Vestibular Rehabiliation Therapy
Other: Conventional treatment — Standing balance training, weight shifting training, walking training, muscle strength training, step-up-and-down training.
  Arms: Conventional Treatment

SUMMARY:
The objective of the study is to determine the effects of stroke conventional therapy compared with the effects of vestibular rehabilitation therapy on balance and post stroke fatigue. The study will be randomized control trial including 2 experimental groups with estimated 28 individual in each group

DETAILED DESCRIPTION:
Stroke is the sudden onset of neurological disorders caused by damage to the cerebrovascular arteries. Vascular injury to the brain can be caused by rapid changes in blood pressure and oxygen shortage, resulting in the death of brain cells. Ischemia accounts for 80% of all strokes. Every year, 15 million individuals worldwide suffer from strokes, and five million become permanently disabled. Stroke prevalence is 1.2% in the province of KPK. Over the last 30 years, the burden caused by stroke has significantly increased, and it has become one of the most common causes of mortality globally. . The central nervous system's sensory (visual, vestibular, somatosensory) and motor systems work together to maintain balance. Patients who have had a stroke are more likely to fall than healthy people due to a variety of impairments in motor and cognitive processes. Vestibular dysfunction may potentially cause falls in this patient population due to poor postural control. It has been found that post stroke patients are more prone than healthy controls to lose standing postural stability under vestibular stimulation. Fatigue is a common post stroke consequence, with a prevalence of between 16 to 74% , and it is considered one of the signs of post stroke depression. However, the fact that patients without depression often complain of fatigue needs a study of "post stroke fatigue" (PSF) as a specific syndrome. This type of fatigue is chronic which can be the only symptom in stroke patients even with adequate neurologic recovery and persists for many years .Fatigue constitutes one of the most common symptoms after a stroke and an important predictor for mortality following stroke. PSF correlates with functional limitations and participation limitations in activities of daily living (ADL), leading to a lower quality of life. Vestibular functions requiring central integration correlate more strongly with fatigue, balance, and walking capacity. Stroke patients have shown an improvement in gait performance, balance, and self-perceived health with vestibular rehabilitation. It has been demonstrated that vestibular therapy has greater benefits on gait in stroke patients. Vestibular rehabilitation therapy (VRT) promote gaze stability, improve postural stability and facilitate sensory integration for patients. VRT was found to be beneficial for improving balance in patients with peripheral vestibular impairment. Cawthorne and Cooksey Exercise Program refers to Vestibular Rehabilitation Therapy. They are exercises that gradually train the eye and body muscles to use visual and proprioceptive signals to compensate for missing or disturbed vestibular signals (which cause poor balance and coordination).Gaze stabilization exercises (GSEs), a type of vestibular therapy, including substitution and adaptation exercises that use the vestibulo-ocular reflex (VOR). Substitution exercises are designed to promote different approaches (saccadic eye movement and smooth tracking activities) to compensate for inadequate vestibular function. Adaptation exercises are long-term alterations in the neural response to head motions that aim to reduce symptoms and normalize gaze and postural stability. GSEs can improve the balance function, confidence, and cognition in older adults with mild cognitive dysfunction .VOR gain has a certain effect on the balance and posture of people following stroke. Balance is common consequence among post stroke patients and increase the risk of fall. The central nervous system's sensory (visual, vestibular, somatosensory) and motor systems work together to maintain balance and prevalence of post stroke fatigue is between 16 to 74% which is high and also the Vestibular functions having highly significant relation with fatigue, and balance and limited evidence on vestibular rehabilitation on post stroke fatigue. That's why this study aims to assess the effect of vestibular rehabilitation training on balance and post-stroke fatigue

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with stroke.
* Ability to stand for at least 1 minute without support.
* Fatigue Assessment Scale (FAS) score ≥ 24.
* Willingness to participate

Exclusion Criteria :

* Cognitive Impairment.
* Severe unilateral spatial neglect.
* Severe aphasia.
* Patients who are not willing.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-03-21 (Estimated); Study Completion 2025-03-21 (Estimated)

PRIMARY OUTCOMES:
1. Berg Balance Scale | 8 weeks
  changes from the baseline, Berg balance scale (BBS) is used for assessment of balance and fall risk, Higher scores on the BBS indicate greater independence and better ability to balance. In contrast, lower scores indicate a greater fall risk Items DESCRIPTION SCORE (0-4) Sitting to standing, Standing unsupported, Sitting unsupported, Standing to sitting, Transfers , Standing with eyes closed , Standing with feet together, Reaching forward with outstretched arm, Retrieving object from floor, Turning to look behind, Turning 360 degrees, Placing alternate foot on stool, Standing with one foot in front, Standing on one foot, TOTAL __/56
Fatigue Assessment Scale | 8 weeks
  The FAS questionnaire was used to assess fatigue symptoms. This self-report questionnaire includes 10 items based on Likert's 5-point scale (1 = never, 5 = often). FAS scores vary from 10 to 50, with higher scores indicating increased fatigue. Fatigue in stroke patients was set at 24 based on the FAS. Total score range from 10 to 50. less than 22 indicates normal, 22 to 34 indicate mild to moderate fatigue,35 or more indicate severe fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Azhar MS-NMPT, Principal Investigator — Riphah International University
Locations (1):
- Helping Hand Institute of rehabilitation, Mānsehra, Khyber Pakhtunkhuwa, Pakistan

IPD SHARING:
Plan to Share IPD: No